CLINICAL TRIAL: NCT02928237
Title: Effect of the Transcranial Direct Current Stimulation (tDCS) of the Motor Cortex on Chronic Abdominal Pain in Patients With Hepatocellular Carcinoma
Brief Title: Effect of tDCS on Chronic Abdominal Visceral Pain in HCC Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Mohamed Abdelhameed, Resident at Anaesthesia, ICU and pain management department,Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 481186
Record Dates: First submitted 2016-03-26; First posted 2016-10-10 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Abdominal Pain
Keywords: tDCS; cancer liver; chronic abdominal pain; VAS; VDS; HAM-D; BPI; analgesia
MeSH Terms: conditions — Abdominal Pain; Carcinoma, Hepatocellular; Agnosia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Real tDCS (Active Comparator): In the active stimulation condition a constant current of active transcranial direct current stimulation (tDCS) of 2mA intensity was applied for 30 minutes,over primary motor cortex M1. The treatment was repeated every day for 10 consecutive days.
  Interventions: Device: transcranial direct current stimulation tDCS
- Sham tDCS (Placebo Comparator): Sham tDCS was applied using the same parameters but only for 30 seconds then the machine is deactivated.
  Interventions: Device: transcranial direct current stimulation tDCS

INTERVENTIONS:
Device: transcranial direct current stimulation tDCS — A battery driven DC stimulator (neuroConn Gmbh,98693 llmenau, Germany)

SUMMARY:
To evaluate the effect of transcranial direct current stimulation (tDCS) applied to the motor cortex to reduce chronic abdominal visceral pain in a group of participants with hepatocellular carcinoma

DETAILED DESCRIPTION:
This study will be carried out in Assiut University Hospital pain clinic and in participation of department of neuropsychiatry in Assiut University Hospital. After obtaining approval of hospital ethical committee, informed written consent will be taken from all patients with malignant visceral pain to be involved in this study.

In these study investigators test the hypothesis that Does transcranial direct current stimulation induce analgesia in chronic abdominal visceral pain due to liver cancer ?

Preparation:

The patient will seat in a comfortable chair and will be asked to relax as much as possible. tDCS was delivered using a battery driven DC stimulator (neuroConn Gmbh,98693 llmenau, Germany). Current was delivered by electrodes encased in sponge pads soaked with 1% saline solution. The machine was kept behind the participant and out of their view at all times. For both the active and sham conditions, the anode was placed over the motor cortex of the patient and the cathode was placed over the contralateral supraorbital region. Electrodes were secured using soft elastic straps.

In the active stimulation condition a constant current of 2mA intensity was applied for 30 minutes with a 5-second ramp phase at the beginning. In the sham stimulation condition the machine was activated for 30 seconds using identical parameters but was then switched off without the patient's knowledge. This sham control is commonly employed because over the initial 30 seconds of stimulation, an initial sensation of tingling under the electrode fades away. Patients are less likely to distinguish active from sham conditions if the initial period of tingling is present in both.

Patients were evaluated by verbal descriptor scale (VDS), visual analog scale (VAS), and Hamilton rating scale for depression (HAM-D) at the baseline, after 1st, 5th, 10th session, and 1 month after end of sessions.

ELIGIBILITY:
Inclusion Criteria:

* All patients of above 18 years old, with malignant visceral pain due to primary liver cancer or on top of cirrhosis, resistant to medical treatment for at least 2 months or associated with significant adverse effect from medication will be involved in this study

Exclusion Criteria:

* Investigators will exclude patients with intracranial metallic devices or with pacemakers or any other device. Investigators also exclude those with extensive myocardial ischemia and those known to have epilepsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-04; Primary Completion 2016-04 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
visual analog scale (VAS) | one month
  measurement of reduction of chronic abdominal pain in cancer liver patients.
verbal descriptor scale (VDS) | one month
  measurement of reduction of chronic abdominal pain in cancer liver patients.

SECONDARY OUTCOMES:
Hamilton rating scale for depression (HAM-D) | one month
  Measurement of reduction of depression

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Ibrahim NM, Abdelhameed KM, Kamal SMM, Khedr EMH, Kotb HIM. Effect of Transcranial Direct Current Stimulation of the Motor Cortex on Visceral Pain in Patients with Hepatocellular Carcinoma. Pain Med. 2018 Mar 1;19(3):550-560. doi: 10.1093/pm/pnx087. PMID 28605527